CLINICAL TRIAL: NCT04068974
Title: Camrelizumab Combined With Apatinib for Recurrent Platinum-resistant Ovarian Cancer: a Phase 2 Single-arm Prospective Study
Brief Title: Camrelizumab /Apatinib for Recurrent Platinum-resistant Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lingya Pan, Chief, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-OvaC-IIT-SHR1210-APA
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Recurrent Platinum-resistant Ovarian Cancer
Keywords: Ovarian Cancer; Recurrent Platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Camrelizumab (SHR-1210) 200mg, once every 2 weeks, each 4 weeks is 1cycle. Apatinib :250 mg po qd
  Interventions: Drug: Camrelizumab (SHR-1210); Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab (SHR-1210) — Anticancer T-cell activity is regulated by multiple suppressive mechanisms, including tumour-expressed programmed cell death ligand 1 (PD-L1) signalling to the T-cell inhibitory receptor (programmed death protein 1 [PD-1]). Monoclonal antibodies like SHR-1210 that can block this pathway.
Drug: Apatinib — Apatinib is an oral small-molecule tyrosine kinase inhibitor that selectively binds to and inhibits VEGF receptor 2.

SUMMARY:
This study is intend to improve the progression-free survial of the recurrent paltinum-resistant ovarian cancer. All the participants will receive camrelizumab combined with apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent -resistant epithelial ovarian cancer, fallopian tube cancer and primary peritoneal cancer previously received twice or more platinum chemotherapy before enrolment;
2. Recurrence occurred within 6 months after the last platinum-containing chemotherapy and had experienced at least one platinum-sensitive recurrent in the past.;
3. Aged 18-70 years;
4. An Eastern Cooperative Oncology Group performance status of 0-2;
5. According to the solid tumor efficacy evaluation standard (RECIST1.1) or i RECIST, at least one measurable lesion, with maximum diameter > 1 cm and lymph node metastasis > 1.5 cm, and the target lesion is not suitable for surgical treatment; the target lesion has not received radiotherapy or recurred in the field of radiotherapy.
6. Expected survival ≥ 4 months;
7. The function of vital organs meets the following requirements： Hemoglobin≥80g/L; Absolute neutrophil count≥1.5*109/L；Platelets≥100

   *109/L; Creatinine≤1.5 times ULN; Urea nitrogen≤2.5 times ULN; Total Bilirubin≤ULN; ALT and AST ≤ 2.5 times ULN; Albumin≥25g/L; TSH≤ULN(if TSH is abnormal, normal T3 and T4 also can acceptable)
8. The subject should be aware of the purpose of the study and the operations required by the study and volunteer to participate in the study before sign the informed consent form.

Exclusion Criteria:

1. Primary platinum refractory patients (first platinum-containing chemotherapy with recurrence within 6 months)
2. Previously exposed to other anti-angiogenic small-molecule TKI drugs, such as pazopanib, sorafenib, regorafenib, cilnitraz, etc. or anti-angiogenic mAbs such as bevacizumab ; or had used an anti-PD-1 antibody, an anti-CTLA-4 antibody, TCR-T, CAR-T and other immune therapy; or 4 weeks before the first administration participated in any other clinical trials of anticancer drugs; or before the first dose Live attenuated vaccines are accepted within 4 weeks or during the study period.
3. Target lesions observed received radiotherapy
4. Other malignant tumors have occurred in the past 3 years..
5. Immunosuppressive drugs used within 14 days prior to the first use of SHR-1210, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (ie, no more than 10 mg/day of turmeric or equivalent drug physiological dose) Other corticosteroids).
6. Late-stage patients with symptomatic, disseminated to visceral, short-term risk of life-threatening complications (including uncontrolled large amounts of exudate [thoracic, pericardium, abdominal cavity], pulmonary lymphangitis, and more than 30% liver involvement patients).
7. Any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, decreased thyroid function; subjects with vitiligo or complete remission asthma in childhood and without any intervention, all above can be included; asthma requiring medical intervention for bronchodilators should be excluded).

8 Metastatic foci of the central nervous system have significant symptoms, such as headache, cerebral edema and blurred vision 9. CT or MRI showed tumor lesion 5mm away from the great blood vessel, or tumor invading the local great blood vessel, or accompanied by tumor thrombus formation of the great vein (inferior vena cava of iliac vessel, superior vena cava of pulmonary static vein) 10. Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite with the optimal medical treatment.

11. Grade II or higher myocardial ischemia, myocardial infarction or poor control arrhythmia (including male with QTc interval ≥ 450ms, or female with QTc interval≥ 470ms). According to NYHA criteria, grade III to IV cardiac insufficiency, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%; myocardial infarction occurred within 6 months before enrollment, New York Heart Association Level II or above failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, pericardial disease with clinically significant, or electrocardiogram suggesting acute ischemia or abnormal active conduction system.

12, Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5ULN), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy.

13. Half of a teaspoons (2.5 ml) or more hemoptysis was found within the first 2 months or there were significant clinical bleeding symptoms or clearly propensity bleeding within 3 months before participant in the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ or above in baseline or vasculitis; artery or venous thrombosis events within 6 months prior to the study, such as cerebrovascular accidents (Including transient ischemic attacks, cerebral hemorrhage, cerebral infarction, deep vein thrombosis and pulmonary embolism.

14. Severe infections within 4 weeks prior to accept medication (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever during screening/first administration >38.5 °C 15. Those who have a history of psychotropic drug abuse and are unable to quit or have mental disorders.

16. Major surgical procedures were performed within 4 weeks before the first administration. Or open wounds or fractures.

17. There are obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction. Or sinus or perforation of empty organs within 6 months.

18. Routine urine test indicated that urinary protein (++) or more, confirmed urinary protein (>1.0 g) within 24 hours.

19. Patients with a history of allergy may be potentially allergic or intolerant to Apatinib and biological agents SHR-1210.

20. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA (> 500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of the analysis method) or co-infection with hepatitis B and hepatitis C.

21. There is any situation that may damage the subject or cause the subject to fail to meet or implement the research requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to two years
  The proportion of participants with tumor size reduction of a predefined amount and for a minimum time period.

SECONDARY OUTCOMES:
Progression Free Survival | Up to two years
  The time from treatment until objective tumor progression or death, whichever occurs first.
Disease Control Rate | Up to two years
  The proportion of patients with complete response, partial response or keep stable diease after accept treatment.
Duration of Response (DoR) | Up to two years
  The time from firstly complete response or partly response to progressive disease.
Assessment of safety | Up to two years
  The quantity and degree of adverse event and serious adverse event from

CONTACTS AND LOCATIONS:
Overall Officials: Pan lingya, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No